CLINICAL TRIAL: NCT04521920
Title: Providing Comprehensive Harm Reduction Via Telemedicine for PWID Using Syringe Services Programs: a Feasibility Study
Brief Title: Providing Suboxone and PrEP Using Telemedicine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00104147; Pro00104148 (Other: Duke University Health System)
Record Dates: First submitted 2020-08-18; First posted 2020-08-21 (Actual); Results first posted 2023-06-08 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Opioid Use; Opioid-use Disorder; Risk Reduction; Hiv
Keywords: opioid; medication for opioid use disorder; syringe services program; telemedicine; PrEP; HIV prevention; retention in care; suboxone; buprenorphine; feasibility; acceptability
MeSH Terms: conditions — Opioid-Related Disorders; Risk Reduction Behavior; Acquired Immunodeficiency Syndrome | interventions — Buprenorphine, Naloxone Drug Combination; Pre-Exposure Prophylaxis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Medication and telemedicine follow up (Experimental): All participants are provided with Suboxone and/or PrEP and follow up visits will be conducted via telemedicine
  Interventions: Drug: Suboxone; Drug: PrEP

INTERVENTIONS:
Drug: Suboxone — Enrolled participants will be prescribed PrEP and/or Suboxone. Follow up visits will be conducted by telemedicine. We are testing whether telemedicine is a feasible method for follow up.
Drug: PrEP — Enrolled participants will be prescribed PrEP and/or Suboxone. Follow up visits will be conducted by telemedicine. We are testing whether telemedicine is a feasible method for follow up.
  Other Names: Pre-Exposure Prophylaxis (PrEP)

SUMMARY:
The purpose of this study is to provide medication for opioid use disorder (MOUD) with buprenorphine and naloxone, or bup/nx, and pre-exposure prophylaxis (PrEP) for HIV prevention for persons who inject opioids accessing syringe services programs (SSPs), as part of a comprehensive harm reduction program, and assess the acceptability and feasibility of using telemedicine to implement the program.

The initial visit will be conducted in person or remotely via telemedicine given COVID-19 protocols at the SSP sites in Charlotte and Wilmington, North Carolina (NC); follow-up visits will be conducted via telemedicine.

DETAILED DESCRIPTION:
The purpose of this study is to provide medication for opioid use disorder (MOUD) with buprenorphine and naloxone, or bup/nx, and pre-exposure prophylaxis (PrEP) for HIV prevention for persons who inject opioids accessing syringe services programs (SSPs), as part of a comprehensive harm reduction program, and assess the acceptability and feasibility of using telemedicine to implement the program.

The study objectives are the following:

1. To assess uptake and persistence to bup/nx and PrEP as part of a comprehensive harm reduction program among people who inject drugs using SSPs.
2. To assess feasibility and acceptability of implementing a telemedicine-based MOUD and PrEP program

The study population is people who inject drugs, specifically opioids, and who access services at SSPs in Charlotte and Wilmington, NC. The study team will enroll 20 PWID accessing the participating SSPs in Charlotte and Wilmington, NC (10 from each site). Participants will be enrolled in the study for 6 months. At the end of the study, they will be referred to MOUD and PrEP providers identified in the community.

Data collection

Enrollment visit:

The study coordinator will administer the SOCRATES 8D and a baseline survey to collect demographics, HIV risk behaviors, and substance use history. Participants will undergo laboratory testing at the SSP to determine eligibility and enrolled participants will be prescribed bup/nx and PrEP free of charge.

Follow up visits:

Follow-up visits will be conducted via telemedicine at the SSPs. For the first month (Month 1), telemedicine visits will be weekly with each study participant to ensure that they are stable on the appropriate bup/nx dose. Starting at Month 2, the telemedicine visits will take place monthly. Participants will be asked to complete a questionnaire at Month 3 and Month 6 which include questions on HIV risk and drug use, as well as adherence evaluation for both bup/nx and PrEP.

By the end of the study, we hope to determine the following:

* The proportion of persons who demonstrate no or minimal opioid use
* The proportion of persons who remain HIV negative.
* Retention or persistence in care

We will also examine whether participants are more apt to remain on paired/combined therapy compared to individual treatment.

Under the secondary ID, IRB Pro00104148, we will conduct an ancillary study to contribute to the overall feasibility purpose of the primary study (Pro00104147) by collecting qualitative data from program users. The ancillary study will include conducting in-depth interviews (IDIs) with 10 to 20 participants in the primary study at the end of their month 1 telemedicine visit and at the end of their month 6 telemedicine visit (completion of the primary study). We will use applied thematic analysis to analyze participants' narratives. We chose to position this assessment within an ancillary protocol rather that embed it within the primary study in order to reduce the potential for socially desirable responses.

ELIGIBILITY:
Inclusion Criteria:

* History of self-report injection opioid use in the past 6 months
* Participate in SSPs,
* HIV negative
* Willing to take bup/nx and PrEP for 6 months
* No medical contraindications for these medications
* Not pregnant
* 18 years or older
* Not currently taking PrEP
* Not currently taking any form of MOUD
* History of sharing injection or drug preparation equipment or risk of sexual acquisition of HIV (such as engaging in sex work or men who have sex with men) in the past 6 months

Exclusion Criteria:

* Positive pregnancy test including during the course of the study
* Positive HIV test at enrollment
* Altered mental status in which participant cannot sign a consent form
* Renal insufficiency/failure
* Hepatitis B surface antigen positive
* Becoming incarcerated during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehri McKellar, MD, Principal Investigator — Duke Health
Locations (3):
- United States (3):
  - Queen City Needle Exchnge, Charlotte, North Carolina
  - Duke Department of Population Health Sciences, Durham, North Carolina
  - North Carolina Harm Reduction Coalition, Wilmington, North Carolina

IPD SHARING:
Plan to Share IPD: No
We will not share IPD with other researchers.

REFERENCES:
- [Background] Mars SG, Bourgois P, Karandinos G, Montero F, Ciccarone D. "Every 'never' I ever said came true": transitions from opioid pills to heroin injecting. Int J Drug Policy. 2014 Mar;25(2):257-66. doi: 10.1016/j.drugpo.2013.10.004. Epub 2013 Oct 19. PMID 24238956
- [Background] Lankenau SE, Teti M, Silva K, Jackson Bloom J, Harocopos A, Treese M. Initiation into prescription opioid misuse amongst young injection drug users. Int J Drug Policy. 2012 Jan;23(1):37-44. doi: 10.1016/j.drugpo.2011.05.014. Epub 2011 Jun 20. PMID 21689917
- [Background] Young AM, Havens JR. Transition from first illicit drug use to first injection drug use among rural Appalachian drug users: a cross-sectional comparison and retrospective survival analysis. Addiction. 2012 Mar;107(3):587-96. doi: 10.1111/j.1360-0443.2011.03635.x. Epub 2011 Oct 26. PMID 21883604
- [Background] Al-Tayyib AA, Rice E, Rhoades H, Riggs P. Association between prescription drug misuse and injection among runaway and homeless youth. Drug Alcohol Depend. 2014 Jan 1;134:406-409. doi: 10.1016/j.drugalcdep.2013.10.027. Epub 2013 Nov 7. PMID 24300900
- [Background] Valdez A, Neaigus A, Cepeda A. Potential risk factors for injecting among Mexican American non-injecting heroin users. J Ethn Subst Abuse. 2007;6(2):49-73. doi: 10.1300/J233v06n02_05. PMID 18192204
- [Background] Choopanya K, Martin M, Suntharasamai P, Sangkum U, Mock PA, Leethochawalit M, Chiamwongpaet S, Kitisin P, Natrujirote P, Kittimunkong S, Chuachoowong R, Gvetadze RJ, McNicholl JM, Paxton LA, Curlin ME, Hendrix CW, Vanichseni S; Bangkok Tenofovir Study Group. Antiretroviral prophylaxis for HIV infection in injecting drug users in Bangkok, Thailand (the Bangkok Tenofovir Study): a randomised, double-blind, placebo-controlled phase 3 trial. Lancet. 2013 Jun 15;381(9883):2083-90. doi: 10.1016/S0140-6736(13)61127-7. Epub 2013 Jun 13. PMID 23769234
- [Background] Velander JR. Suboxone: Rationale, Science, Misconceptions. Ochsner J. 2018 Spring;18(1):23-29. No abstract available. PMID 29559865
- [Background] Sullivan LE, Moore BA, Chawarski MC, Pantalon MV, Barry D, O'Connor PG, Schottenfeld RS, Fiellin DA. Buprenorphine/naloxone treatment in primary care is associated with decreased human immunodeficiency virus risk behaviors. J Subst Abuse Treat. 2008 Jul;35(1):87-92. doi: 10.1016/j.jsat.2007.08.004. Epub 2007 Oct 15. PMID 17933486
- [Background] Bazzi AR, Biancarelli DL, Childs E, Drainoni ML, Edeza A, Salhaney P, Mimiaga MJ, Biello KB. Limited Knowledge and Mixed Interest in Pre-Exposure Prophylaxis for HIV Prevention Among People Who Inject Drugs. AIDS Patient Care STDS. 2018 Dec;32(12):529-537. doi: 10.1089/apc.2018.0126. Epub 2018 Oct 11. PMID 30311777
- [Background] Edelman EJ, Moore BA, Calabrese SK, Berkenblit G, Cunningham C, Patel V, Phillips K, Tetrault JM, Shah M, Fiellin DA, Blackstock O. Primary Care Physicians' Willingness to Prescribe HIV Pre-exposure Prophylaxis for People who Inject Drugs. AIDS Behav. 2017 Apr;21(4):1025-1033. doi: 10.1007/s10461-016-1612-6. PMID 27896552
- [Background] Molfenter T, Fitzgerald M, Jacobson N, McCarty D, Quanbeck A, Zehner M. Barriers to Buprenorphine Expansion in Ohio: A Time-Elapsed Qualitative Study. J Psychoactive Drugs. 2019 Jul-Aug;51(3):272-279. doi: 10.1080/02791072.2019.1566583. Epub 2019 Feb 7. PMID 30732542
- [Background] Haffajee RL, Lin LA, Bohnert ASB, Goldstick JE. Characteristics of US Counties With High Opioid Overdose Mortality and Low Capacity to Deliver Medications for Opioid Use Disorder. JAMA Netw Open. 2019 Jun 5;2(6):e196373. doi: 10.1001/jamanetworkopen.2019.6373. PMID 31251376
- [Background] Zheng W, Nickasch M, Lander L, Wen S, Xiao M, Marshalek P, Dix E, Sullivan C. Treatment Outcome Comparison Between Telepsychiatry and Face-to-face Buprenorphine Medication-assisted Treatment for Opioid Use Disorder: A 2-Year Retrospective Data Analysis. J Addict Med. 2017 Mar/Apr;11(2):138-144. doi: 10.1097/ADM.0000000000000287. PMID 28107210
- [Background] Weintraub E, Greenblatt AD, Chang J, Himelhoch S, Welsh C. Expanding access to buprenorphine treatment in rural areas with the use of telemedicine. Am J Addict. 2018 Dec;27(8):612-617. doi: 10.1111/ajad.12805. Epub 2018 Sep 28. PMID 30265425
- [Background] Centers for Disease Control and Prevention. Revised guidelines for HIV counseling, testing, and referral. MMWR Recomm Rep. 2001 Nov 9;50(RR-19):1-57; quiz CE1-19a1-CE6-19a1. PMID 11718472
- [Derived] McKellar MS, Des Marais AC, Chen H, Choi Y, Lilly R, Ayers D, Bennett J, Kestner L, Perry B, Poley S, Corneli A, Meade CS, Sachdeva N. Providing medication for opioid use disorder and HIV pre-exposure prophylaxis at syringe services programs via telemedicine: a pilot study. Harm Reduct J. 2024 Mar 26;21(1):69. doi: 10.1186/s12954-024-00983-2. PMID 38532395
- [Derived] Corneli A, Perry B, Des Marais A, Choi Y, Chen H, Lilly R, Ayers D, Bennett J, Kestner L, Meade CS, Sachdeva N, McKellar MS. Participant perceptions on the acceptability and feasibility of a telemedicine-based HIV PrEP and buprenorphine/naloxone program embedded within syringe services programs: a qualitative descriptive evaluation. Harm Reduct J. 2022 Dec 3;19(1):132. doi: 10.1186/s12954-022-00718-1. PMID 36463214

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited people who inject drugs, who access services at syringe services programs in Wilmington and Charlotte, North Carolina.
Period: Overall Study
Arm/Group | Medication and Telemedicine Follow up
Started | 17
Month 3 | 13
Completed | 12
Not Completed | 5

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Arm/Group | Medication and Telemedicine Follow up
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 17
Education [Count of Participants; unit: Participants] — Education completed measured via self-report
  Participants
    Some high school | 3
    High school or GED | 4
    Any college | 10
Insurance status [Count of Participants; unit: Participants] — Insurance coverage measured via self-report
  Participants
    Private | 3
    Public | 1
    No insurance | 13
Relationship status [Count of Participants; unit: Participants] — Relationship status measured via self-report
  Participants
    Single/ Separated | 11
    Married/ Partnered | 6
Employment [Count of Participants; unit: Participants] — Employment status measured via self-report
  Participants
    Working full-time | 3
    Working part-time | 5
    Student | 1
    Disabled, unable to work | 1
    Unemployed | 6
    Stay at home parent | 1
Ever taken Suboxone [Count of Participants; unit: Participants] — Whether the participant has ever taken Suboxone prior to the study measured via self-report
  Participants
    Yes | 16
    No | 1
Ever Overdosed [Count of Participants; unit: Participants] — Whether the participant has ever overdosed on heroin, fentanyl, or prescription pain medication measured via self-report
  Participants
    Yes | 9
    No | 8
Access to technology [Number; unit: participants] — Technology participants have access to measured via self-report
  participants
    Computer with video camera | 6
    Computer without video camera | 1
    Smartphone | 17
    Tablet | 1
    Basic telephone (without internet capabilities) | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Demonstrate no or Minimal Opioid Use at 3 Months
Description: Defined as self-reported opioid use in prior month
Time Frame: 3 months
Population: Data not collected on 8 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Medication and Telemedicine Follow up
Number analyzed (Participants) | 9
Participants | 6

2. Primary Outcome: Number of Participants Who Demonstrate no or Minimal Opioid Use at 6 Months
Description: Defined as self-reported opioid use in prior month.
Time Frame: 6 months
Population: Data not collected on 11 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Medication and Telemedicine Follow up
Number analyzed (Participants) | 6
Participants | 5

3. Primary Outcome: Number of Participants Who Remain HIV Negative at 3 Months
Description: Measured via negative HIV test.
Time Frame: 3 months
Population: Received labs to confirm HIV status from 8 participants at month 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Medication and Telemedicine Follow up
Number analyzed (Participants) | 8
Participants | 8

4. Primary Outcome: Number of Participants Who Remain HIV Negative at 6 Months
Description: Measured via negative HIV test.
Time Frame: 6 months
Population: Received labs to confirm HIV status from 3 participants at month 6
Measure: Count of Participants; unit: Participants
Arm/Group | Medication and Telemedicine Follow up
Number analyzed (Participants) | 3
Participants | 3

5. Primary Outcome: Persistence in Care at 3 Months
Description: Defined as the number of participants who remain on treatment (MOUD or PrEP).
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Medication and Telemedicine Follow up
Number analyzed (Participants) | 17
Participants | 13

6. Primary Outcome: Persistence in Care at 6 Months
Description: Defined as the number of participants who remain on treatment (MOUD or PrEP).
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Medication and Telemedicine Follow up
Number analyzed (Participants) | 17
Participants | 12

7. Other Pre Specified Outcome: Motivators and Barriers Affecting Medication Adherence and Persistence
Description: Exploratory method, conducted in the form of individual interviews to document the personal experiences and opinions of each participant over time (qualitative method)
Time Frame: 6 month
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Motivators and Barriers Affecting Program Persistence
Description: as for outcome 7
Time Frame: 6 month
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Participant Perceived Usefulness of the Program
Description: as for outcome 7
Time Frame: 6 month
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Participant Perceived Usefulness of the Program
Description: Exploratory method, conducted in the form of individual interviews to document the personal experiences and opinions of each participant (qualitative method)
Time Frame: 1 month
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Participant Satisfaction With the Program
Description: as for outcome 7
Time Frame: 6 month
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Participant Satisfaction With the Program
Description: as for outcome 10
Time Frame: 1 month
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Perceptions of Medical Care Quality Via a Telemedicine Video Platform
Description: Exploratory method, conducted in the form of individual interviews to document the personal experiences of each participant (qualitative method)
Time Frame: 6 month
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Ease/Difficulty of Accessing the Telemedicine Video Platform
Description: as for outcome 13
Time Frame: 1 month
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Ease/Difficulty of Visiting a SSP to Meet With a Provider Via Telemedicine
Description: Exploratory method, conducted in the form of individual interviews to document the personal experiences of each participant over time (qualitative method)
Time Frame: 6 month
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Ease/Difficulty of Visiting a SSP to Meet With a Provider Via Telemedicine
Description: as for outcome 13
Time Frame: 1 month
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 6 months
Arm/Group | Medication and Telemedicine Follow up
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-19): https://cdn.clinicaltrials.gov/large-docs/20/NCT04521920/Prot_SAP_000.pdf